CLINICAL TRIAL: NCT04165213
Title: A Training and Fidelity Model to Move and Scale Evidence-based Dementia Care and Caregiver Support Programs Into Practice: The Case for COPE in PACE Service Settings
Brief Title: Care of Persons With Dementia in Their Environments (COPE) in Programs of All-Inclusive Care of the Elderly (PACE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Drexel University (Other); Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 831688
Record Dates: First submitted 2019-08-26; First posted 2019-11-15 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Frontotemporal Dementia; Dementia; Multi-Infarct Dementia; Vascular Dementia; Mixed Dementia; Alzheimer Disease; Lewy Body Disease; Pick Disease; Neurocognitive Disorders
MeSH Terms: conditions — Frontotemporal Dementia; Dementia; Dementia, Multi-Infarct; Dementia, Vascular; Mixed Dementias; Alzheimer Disease; Lewy Body Disease; Pick Disease of the Brain; Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Instructor-trained COPE clinicians (No Intervention): Clinicians from PACE sites randomized to this study arm (control) will receive instructor-led training in the evidence-based dementia care program called COPE. After clinician consent and enrollment, outcome measures will be collected prior to training (pre-training baseline), after training (post-training baseline), and after delivering COPE to dyads (4 months post-implementation).
  Dyads (caregivers and PLWDs) receiving COPE from Instructor-trained COPE clinicians are represented in the study arms "Caregivers receiving COPE from instructor-trained COPE clinicians" and "PLWDs COPE from instructor-trained COPE clinicians."
  These participants are receiving the usual instructor-led training - not the experimental training.
- COPE module-trained clinicians (Experimental): Clinicians from PACE sites randomized to this study arm (intervention) will receive self-paced online module training in the evidence-based dementia care program called COPE. After clinician consent and enrollment, outcome measures will be collected prior to training (pre-training baseline), after training (post-training baseline), and after delivering COPE to dyads (4 months post-implementation).
  Dyads (caregivers and PLWDs) receiving COPE from module-trained COPE clinicians are represented in the study arms "Caregivers receiving COPE from module-trained COPE clinicians" and "PLWDs COPE from module-trained COPE clinicians."
  Interventions: Behavioral: Care of Older Persons in their Environment (COPE) online module training
- Caregivers receiving COPE from instructor-trained COPE clinicians (No Intervention): Caregivers of eligible PLWDS enrolled at PACE sites randomized to the control arm will be recruited by "instructor-trained COPE clinicians." After initial recruitment, the study team will carry out consent and screening procedures with caregivers and collect caregiver outcome data at baseline (before meeting with COPE clinicians) and follow-up (4 months post-implementation). Caregivers must complete a minimal dose of 4 sessions out of 10 to be included in follow-up measures. Outcomes will be reviewed for change from baseline to follow-up and compared to "caregivers receiving COPE from module-trained COPE clinicians" for non-inferiority.
  These participants are receiving COPE from clinicians trained in the instructor-led COPE training.
- Caregivers receiving COPE from module-trained COPE clinicians (Experimental): Primary caregivers of eligible PLWDS enrolled at PACE sites randomized to the intervention arm will be recruited by "module-trained COPE clinicians." After initial recruitment, the study team will carry out consent and screening procedures with caregivers and collect caregiver outcome data at baseline (before meeting with COPE clinicians) and follow-up (4 months post-implementation). Caregivers must complete a minimal dose of 4 sessions out of 10 to be included in follow-up measures. Outcomes will be reviewed for change from baseline to follow-up and compared to "caregivers receiving COPE from instructor-trained COPE clinicians" for non-inferiority.
  Interventions: Behavioral: Care of Older Persons in their Environment (COPE) online module training
- PLWDs receiving COPE from instructor-trained COPE clinicians (No Intervention): Eligible PLWDS enrolled at PACE sites randomized to the control arm will be screened for eligibility and initial interest by "instructor-trained COPE clinicians" before caregiver recruitment. PLWDs will only be enrolled if caregivers consent to participate. PLWD outcome data will be collected at baseline (before meeting with COPE clinicians) and follow-up (4 months post-implementation). A minimal dose of 4 sessions out of 10 sessions must be completed for PLWD to be included in follow-up measures. Outcomes will be reviewed for change from baseline to follow-up and compared to "PLWDS receiving COPE from module-trained COPE clinicians" for non-inferiority.
  These participants are receiving COPE from clinicians trained in the usual instructor-led COPE training.
- PLWDs receiving COPE from module-trained COPE clinicians (Experimental): Eligible PLWDS enrolled at PACE sites randomized to the intervention arm will be screened for eligibility and initial interest by "module-trained COPE clinicians" before caregiver recruitment. PLWDs will only be enrolled if caregivers consent to participate. PLWD outcome data will be collected at baseline (before meeting with COPE clinicians) and follow-up (4 months post-implementation). A minimal dose of 4 sessions out of 10 sessions must be completed for PLWD to be included in follow-up measures. Outcomes will be reviewed for change from baseline to follow-up and compared to "PLWDS receiving COPE from instructor-trained COPE clinicians" for non-inferiority.
  Interventions: Behavioral: Care of Older Persons in their Environment (COPE) online module training

INTERVENTIONS:
Behavioral: Care of Older Persons in their Environment (COPE) online module training — An online module version of training for clinicians (OTs and RNs) in the evidence-based dementia caregiving program called Care of Older Persons in their Environment (COPE) is the intervention being tested for non-inferiority against the usual instructor-led COPE training. COPE modules include rich multimedia content, simulated scenarios, interactive assessments to keep the learner engaged The content is packaged into the latest the latest Shareable Content Object Reference Model (SCORM) specifications, which will allow for repurposing and sharing with other institutions. Each of the ten modules last 45-60 minutes.
  Other Names: COPE online training
  Arms: COPE module-trained clinicians; Caregivers receiving COPE from module-trained COPE clinicians; PLWDs receiving COPE from module-trained COPE clinicians

SUMMARY:
The protocol is organized into three Phases - In Phase I an online training program will be developed in "Care of Persons with Dementia in their Environments" (COPE) -an evidence-based bio-behavioral dementia program -using state-of-the science simulation and best online learning practices. In addition an automated approach to fidelity monitoring using computational linguistics (automatic classification programs) will be developed. In Phase II, ten long term care community-based (PACE) organizations will be randomized into two groups; 5 PACE organizations will serve as the "control" site in which staff training will be provided via the traditional high intensity face-to-face training in the COPE program. 5 PACE organizations will serve as the comparison and staff will be trained using the online COPE training program. Phase II will evaluate the whether an online training program is the same or better in improving PACE staff competency and fidelity to COPE principles and protocols compared to a high intensity face-to-face traditional form of training. In Phase III the efficacy of the COPE program on PACE participant outcomes by type of COPE training will be evaluated. Each of the PACE organizations will enroll 5 persons with dementia and their caregivers in the study. This will yield 50 family dyads (25 dyads in traditional training sites and 25 dyads in online training sites). Dyads will be followed for 4 months. Non-inferiority analysis will be used to assess whether dyads will yield the same or better outcomes regardless of how PACE staff were trained.

DETAILED DESCRIPTION:
PHASE 1a - The Online Training Program - We will develop ten self-paced online learning modules. These modules will enable OTs and RNs to participant to have anytime/anywhere access to content and activities to aid their learning. The modules will include rich multimedia content and interactive assessments to keep the learner engaged. The modules will allow for easy packaging of the content into the latest interoperability standards for such content including the latest Shareable Content Object Reference Model (SCORM) specifications, which will allow for repurposing and sharing with other institutions.

To accommodate diversity of learning needs, the modules will be designed using a hyperlearning model with four dimensions. The general principles will begin with the module learning objectives and follow with a review of core concepts and required and/or self-directed learning activities. The mini-lecture component of the modules will include information on the major concepts of the module. Since the modules will be self-paced, the learner can take his/her time going through them and perform in the embedded interactive learning activities. The clinical reasoning dimension will provide the learner with an opportunity for problem-solving and clinical decision-making. This dimension will contain vignettes and case studies with questions requiring analysis and synthesis. The final dimension will be evaluation/ assessment of learning outcomes. This dimension will use teacher-made and standardized pre-and post-tests to assess attainment of specified learning outcomes. The self-paced modules will be highly interactive featuring integrated multimedia content, assessments, and learner evaluations to allow PACE staff to engage with the content at a high level and practice application in simulated scenarios. Each module will require approximately 45-60 minutes/module for the learner to complete. Participants can use the modules separately at different times throughout a training curriculum or they can be assigned at the beginning of a training time by having this information front-loaded.

To develop the modules, we will work intensely in year 01 with an instructional design team at Drexel University with specialists in dementia care, the COPE program and experts in simulation, use of standardized patients, and training of nurses and other health professionals from Penn, Trinity Health and Jefferson. We anticipate the modules to contain the following content: module 1 - introduction to COPE program, research evidence, and core principles underlying the program; module 2 - overview of delivery characteristics, role of RN and OT, three phases (assessment, implementation, generalizability) of the COPE program, permissible adaptations; module 3 and 4-assessment phase, introduction to clinical interview and all assessments and forms; module 5 and 6- implementation phase including helping caregiver identify 3 problem areas, engaging in problem solving and brainstorming, developing and providing an assessment report and offering prescriptions (strategies) for each identified problem area; module 7 and 8 - generalizability phase or helping caregivers use strategies for one problem area to address another and planning for the future; module 9- developing rapport and working with family caregivers from different backgrounds, cultures, living environments and relationships and helping families balance caregiving with other life roles, adjusting approach by level of readiness; module 10 - challenging cases, motivational interviewing, how to explain the program, how to meet caregivers where they are at and provide validation and support.

Scripts for each module will be developed and shared with OTs/RNs who are not part of the study but work within Trinity PACE programs. This will allow for continuous feedback loops to assure that the scenarios meet the needs of PACE staff. We will compare the online program to our traditional 3-day face-to-face training currently used with COPE.

The 3-day training program will be conducted by Dr. Piersol using a slide deck and case presentations as we have previously done. The comparison of the two training programs is described in Phase 2 and 3 below.

PHASE 1b -The Fidelity Monitoring Program- We seek to develop a scalable approach to assess fidelity to the COPE Program when it is implemented in a real-world setting such as PACE using computational linguistics techniques (e.g. natural language processing). The essence of fidelity to the Core Principles of COPE program will be captured by using automatic classification programs that evaluate both the content that should be included in COPE sessions, and the style of delivery. While automatic classification programs have been applied to measure quality metrics of transcribed narratives in the field of psychotherapy (21), it has not been used to measure other aspects of quality- namely fidelity to evidence-based practices or dementia care and caregiver supportive programs. The development of the automated Fidelity Monitoring Program will occur in three steps and will be carried out by a technical team consisting of an expert in content analysis, Dr. Ani Nenkova, and a consultant expert in speech recognition and prosody, Dr Mari Ostendorf. Co- I Nenkova has worked extensively on automatic summarization, evaluation of automatic summarization and readability and linguistic style. The ultimate goal of our efforts is to develop a system that- given a recording of a COPE delivery session (e.g. in real time immediately after interaction between the clinician and the caregiver)- produces a three-tiered score, indicating if the fidelity was 'excellent', 'acceptable' or 'problematic'. Special emphasis will be given to the accuracy of identifying 'problematic' COPE fidelity which is not fateful to training and may not produce the same desired outcomes as intervention delivered with higher fidelity. First, we will obtain n-best list speech recognition of the COPE interaction . This will help mitigate recognition errors in the next stage. Until recently, audio recording transcription was fraught with challenges particularly in sessions involving two or more speakers. Advances in audio signaling and speech recognition have brought technology for automating language analysis within reach. Recent research has suggested that text based features may be more effective than using audio features alone when classifying fidelity in behavioral research (47). Automatic speech recognition software will be used to transcribe sessions and the resulting words will be used in a text-based model of fidelity. All COPE training, practice and implementation sessions will be audio taped with participant consent. There are several of automatic speech recognition tools that we can use. We will pick the one that best balances accuracy of recognition in our domain and privacy.Once the transcripts are obtained, there are two approaches that we will develop and contrast: (1) comparison with a reference delivery and (2) a supervised classification approach. The first has the advantage of needing only a small number of excellent deliveries and several acceptable deliveries, for each of the seven dimensions, while the other needs a larger set of labeled data but would potentially lead to higher accuracy of prediction.

Comparison or similarity to reference (Steps A and B): Our approach will leverage techniques widely used in the evaluation of automatically produced content, such as machine translation and automatic text summarization. In these applications it is not feasible to track system improvement with human judgments of quality. Instead, most of the progress is measured by computing similarity between a set of sample reference text (i.e. what a 'good' translation or a 'good' summary would be) and the system output. Such automatic evaluation approaches are widely used for machine translation (48) and summarization (49). While there have been some concerns that the automatic measures are not fine enough to distinguish between levels of very good context, these measures show strong ability to distinguish 'very bad' content (50,51), (or poor fidelity) aligns with the needs of our project.

In Step A we will compile 10 examples of 'excellent' COPE fidelity deliveries, with the regions where desired aspects is expressed will be explicitly marked, i.e. marked parts where person-environment fit is discussed, or parts of the interaction where the clinician asks open ended questions or confirms the caregiver understanding of the content. Next, new interactions will be ranked by their similarity with the reference 'excellent' interactions (52). In Step 2 we will identify 'problematic' fidelity deliveries. We will make use of 10 negative examples of 'acceptable' but imperfect deliveries. If the new interaction ranks lower than most of these, it will be considered unacceptable or 'problematic'. Parameters and decision rules will be developed at this step to determine cut-off levels for declaring an interaction problematic.

Determination of "excellent" versus "problematic" fidelity ratings of the audio recordings will be assessed by Drs Hirshman and Renz (who were not the original developers of COPE and thus they offer an independent review) using the COPE Adherence Scale developed for the original clinical trial in order to evaluate the extent to which core treatment principles were implemented effectively. Ratings from the Adherence Scale have been standardized such that 1.00 represents perfect fidelity and 0.00 represent complete non-fidelity. The scale was previously modeled off of the NIH REACH I and II fidelity approach. Findings from the combined fidelity ratings will be used to refine the automated fidelity program into a "best model" to be tested in Step C (53).

Supervised classification (Step C) For this approach, we will need to examine all recorded sessions (600+). We will train a supervised classifier or a regression model to predict the score (1 to 3, corresponding to excellent, acceptable and problematic) of a given interaction. We will experiment with a number of classifiers, including deep learning frameworks and more traditional support vector machine and (logistic) regression models.The resulting final validation set of 100 labeled interactions will serve to finalize the best model for fidelity prediction.

PHASE 2 - Evaluation of Online Training Program in Interventionist Uptake and Fidelity Phase 2 of this study involves a series of activities designed to evaluate the whether an online training program is the same or better in improving interventionist uptake of- and fidelity to- COPE principles and protocols compared to a high intensity face-to-face traditional form of training.

PHASE 3 (Aim 3) - Efficacy of COPE on PACE participant outcomes by type of COPE training.

This aim will be accomplished by evaluating dyad outcomes of the COPE program under the two different training approaches. Following training, each of the PACE organizations will enroll 5 persons with dementia and their caregivers in the study. This will yield 50 family dyads (25 dyads in traditional training sites and 25 dyads in online training sites).

The recruitment plan includes the following goals:

25% recruitment complete by August 1, 2022 50% recruitment complete by October 31, 2022 75% recruitment complete by December 28, 2022 100% recruitment complete by February 28, 2023 Data analysis completed by April 28, 2023

ELIGIBILITY:
Inclusion Criteria:

* Our inclusion criteria are purposively broad to reflect the real world case mix of PACE staff, persons living with dementia and their caregivers using PACE programs. Inclusion Criteria: PACE organization staff will be eligible if they are Occupational Therapists (OTs) or Registered Nurses (RNs) employed full time for more than 1 year at the enrolled PACE site and in good standing . Persons with dementia will be eligible if they: a) are a Trinity PACE participant; b) have a diagnosis of dementia or = four errors on the Mental Status Questionnaire (MSQ, 39), which is updated for each PACE participant every 6 months; (The MSQ threshold of = 4 errors is considered moderate cognitive impairment); c) speaks or understands English. Caregivers are eligible to participate if they: a) have primary responsibility for care of the person with dementia (defined as being the responsible party who enrolled the participant in PACE and who provides hands-on or supervisory assistance with one or more instrumental or daily activities of living); b) speak English; c) have a telephone and are willing to participate in 3 telephone interviews (baseline, 4-and 9 month follow-ups); and d) are 21 years of age or older (male or female). While more than one family member may provide care to the person with dementia and participate in the COPE sessions, we will enroll the family member designated as the responsible party for the purpose of evaluating treatment effects.s in online training sites). At 4 months, study outcomes will be assessed.

Exclusion Criteria:

* Persons with dementia will be excluded if they are a) Diagnosed with schizophrenia or bipolar disorder; b) bedbound and unresponsive; c) participating in a concurrent experimental drug study designed to treat agitation or aggressive behaviors. Dyads are not eligible if: a) they plan to move from the area within 9 months, b) either has been hospitalized >3 times in past year; c) either is in active treatment for a terminal illness or are in hospice; and d) caregiver is involved in other support services/trials. These criteria are designed to minimize attrition and exclude caregivers of relatives at high mortality risk who may not benefit from the COPE Program.

Dyads (PLWDS and CGs) will be excluded from the final sample if they do not complete at least 4 COPE sessions.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Hodgson, PhD RN FAAN, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol paper to be published in Contemporary Clinical Reviews.
Supporting Information: Study Protocol
Time Frame: May 2025
Access Criteria: NIH Manuscript Submission System

REFERENCES:
- [Derived] Hodgson NA, McPhillips MV, Hirschman KB, Summerhayes E, Piersol CV, Gitlin LN. Training to Move an Evidence-based Dementia Caregiver Support Program into Practice: A pragmatic, randomized, non-inferiority trial protocol. Contemp Clin Trials Commun. 2025 Apr 5;45:101478. doi: 10.1016/j.conctc.2025.101478. eCollection 2025 Jun. PMID 40248174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Once at least 10 PACE sites agreed to participate, each site was randomized to the control or intervention groups. Clinicians were enrolled and received the type of training that had already been assigned to their site. Intervention = online module training. Control = Instructor-led training. After training, clinicians and staff enrolled dyads (PLWDs & CGs) to receive COPE. Dyads are assigned to the study arm according to which training their clinician received.
Pre-assignment Details: Prior to assignment, the study team worked with Trinity Health PACE to ensure at least 10 PACE sites would enroll in the study.
Units Other Than Participants: sites
Groups:
- Traditional Training: These sites were randomized to the control group. Clinicians at these sites received the traditional instructor-led training in the COPE program before delivering to dyads enrolled at their sites.
- Module Training: These sites were randomized to the intervention group. Clinicians at these sites received the new module training in the COPE program before delivering to dyads enrolled at their sites.
Period: Clinician Enrollment
Arm/Group | Traditional Training | Module Training
Started | 15; 7 sites | 12; 4 sites
Clinician Training Complete | 12; 7 sites (3 clinicians left the study after baseline measures due to staffing issues, workload and competing priorities. They did not receive training/complete this milestone.) | 12; 4 sites
Post-training Surveys Complete | 12; 7 sites | 12; 4 sites
COPE Delivery Complete | 8; 5 sites (1 clinician did not deliver COPE/complete this milestone. 3 clinicians resigned before this milestone.) | 9; 4 sites (2 clinicians did not deliver COPE/complete this milestone. 1 clinician was terminated before completing this milestone.)
Completed | 8; 5 sites | 9; 4 sites
Not Completed | 7; 2 sites | 3; 0 sites
Not completed — Did not deliver COPE to dyads | 1 | 2
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Termination from site | 0 | 1
Period: Caregiver Enrollment
Arm/Group | Traditional Training | Module Training
Started (This is the start of the caregiver enrollment period. Participants numbers are not related to clinician enrollment numbers above.) | 12; 7 sites | 17; 4 sites
Baseline Measures Collected. | 10; 5 sites (2 caregivers left the study before completing baseline measures.) | 12; 4 sites (5 caregivers left the study before completing baseline measures.)
Minimal Dose of COPE (4 Sessions) Received. | 9; 5 sites (1 caregiver left the study based on the PLWD's physician's decision.) | 8; 4 sites (2 caregivers did not receive COPE. 2 caregivers received less than the minimal dose of COPE to be included in sample.)
Completed | 7; 5 sites (2 caregivers were lost to follow up.) | 7; 4 sites (1 caregiver was lost to follow up.)
Not Completed | 5; 2 sites | 10; 0 sites
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — PLWD entered long term care, no longer eligible | 1 | 0
Not completed — PLWD death | 2 | 0
Not completed — Did not receive minimal dose of COPE | 0 | 4
Period: PLWD Enrollment
Arm/Group | Traditional Training | Module Training
Started | 12; 7 sites | 17; 4 sites
Baseline Measures Collected. | 10; 5 sites (2 PLWDs left the study before caregiver completed baseline measures.) | 12; 4 sites (5 PLWDs left the study before caregivers completing baseline measures.)
Minimal Dose of COPE (4 Sessions) Received. | 9; 5 sites (1 PLWD's physician decided they should leave the study.) | 8; 4 sites (2 PLWD caregivers did not receive COPE. 2 PLWD caregivers received less than the minimal dose of COPE to be included in sample.)
Completed | 7; 5 sites | 7; 4 sites
Not Completed | 5; 2 sites | 10; 0 sites
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Entered long term care, no longer eligible | 1 | 0
Not completed — Death | 2 | 0
Not completed — Did not receive minimal dose of COPE | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- COPE Module-trained Clinicians: Clinicians from PACE sites randomized to this study arm (intervention) will receive self-paced online module training in the evidence-based dementia care program called COPE. After clinician consent and enrollment, outcome measures will be collected prior to training (pre-training baseline), after training (post-training baseline), and after delivering COPE to dyads (4 months post-implementation).
  Dyads (caregivers and PLWDs) receiving COPE from module-trained COPE clinicians are represented in the study arms "Caregivers receiving COPE from module-trained COPE clinicians" and "PLWDs COPE from module-trained COPE clinicians."
  Care of Older Persons in their Environment (COPE) online module training: An online module version of training for clinicians (OTs and RNs) in the evidence-based dementia caregiving program called Care of Older Persons in their Environment (COPE) is the intervention being tested for non-inferiority against the usual instructor-led COPE training. COPE modules include rich multimedia content, simulated scenarios, interactive assessments to keep the learner engaged The content is packaged into the latest the latest Shareable Content Object Reference Model (SCORM) specifications, which will allow for repurposing and sharing with other institutions. Each of the ten modules last 45-60 minutes.
- Total: Total of all reporting groups
Arm/Group | Instructor-trained COPE Clinicians | COPE Module-trained Clinicians | Caregivers Receiving COPE From Instructor-trained COPE Clinicians | Caregivers Receiving COPE From Module-trained COPE Clinicians | PLWDs Receiving COPE From Instructor-trained COPE Clinicians | PLWDs Receiving COPE From Module-trained COPE Clinicians | Total
Number analyzed (Participants) | 12 | 12 | 10 | 12 | 10 | 12 | 68
Age, Continuous [Mean (Full Range); unit: years] — Clinician and Caregiver Ages Population: The age of PLWDS was shared by Trinity Health PACE within a limited data set. The true age of participants aged 89 and older could not be included but only in the category "89 years of age and older."
  years
    Mean Age (Years): number analyzed (Participants) | 12 | 12 | 10 | 12 | 0 | 0 | 46
    Mean Age (Years) | 44 [27 to 65] | 48 [30 to 58] | 56 [39 to 77] | 63 [40 to 89] |  |  | 53 [27 to 89]
Age, Customized [Count of Participants; unit: Participants] — PLWD age categories Population: Clinicians and caregivers mean ages are reported in another measure titles "PLWD age categories."
  Participants
    60-69 years: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 12 | 22
    60-69 years |  |  |  |  | 1 | 1 | 2
    70-79 years: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 12 | 22
    70-79 years |  |  |  |  | 4 | 2 | 6
    80-88 years: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 12 | 22
    80-88 years |  |  |  |  | 4 | 7 | 11
    89 years and older: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 12 | 22
    89 years and older |  |  |  |  | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 10 | 11 | 7 | 6 | 57
  Male | 1 | 0 | 0 | 1 | 3 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 1 | 2 | 1 | 6
  Not Hispanic or Latino | 12 | 12 | 8 | 11 | 8 | 10 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6 | 2 | 7 | 21
  White | 10 | 10 | 5 | 5 | 6 | 4 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 2 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Determinants of Implementation Behavior Questionnaire (Clinicians)
Description: The Determinants of Implementation Behavior Questionnaire (DIBQ) contains 93 items assessing 18 domains and is used to identify determinants of implementation behaviors in order to be able to develop effective strategies to improve healthcare professionals' implementation behaviors. Clinicians in this study were assessed for implementation behavior at post training baseline (prior to COPE implementation) and at follow up (post-implementation) for two DIBQ domains, "knowledge" and "skills." These two domains have demonstrated good discriminant validity and are highly correlated in recent studies (https://doi.org/10.1186/1748-5908-9-33). Participants answer each item with a response from 1 (strongly disagree agree) to 5 (strongly agree) with an option to refuse to respond (score of 0). Each domain has a minimum total score of 0 and maximum total score of 10. Higher scores are positive and indicate improved knowledge and skills in COPE.
Time Frame: Post-training baseline, 14 months
Population: These outcome measures were collected from clinicians in the control and intervention study arms at post-training baseline (just after training) and follow-up (after implementing COPE to dyads). The means reported are change scores between those timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Instructor-trained COPE Clinicians | COPE Module-trained Clinicians
Number analyzed (Participants) | 9 | 8
score on a scale
  Domain 1 (knowledge) change score | 0.06 (0.53) | -0.25 (0.76)
  Domain 2 (skills) change score | 0.33 (0.87) | 0.06 (0.78)

2. Primary Outcome: Perceived Change for Better Index (Caregivers)
Description: The Perceived Change for Better Index is a 13-item scale that measures caregiver appraisals of self-improvement or decline in areas of well-being within a month of survey completion. Caregivers rate items on a 5-point Likert-type scale (1 = became much worse, 2 = became somewhat worse, 3 = stayed the same, 4 = improved somewhat, 5 = improved a lot). Total scores at one time point range from 13-65. Higher scores indicate better outcomes.
Time Frame: Baseline, 4 months
Population: The means reported indicate the change from baseline to follow up. A positive value indicates an improved perception of well being and better outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers Receiving COPE From Instructor-trained COPE Clinicians | Caregivers Receiving COPE From Module-trained COPE Clinicians
Number analyzed (Participants) | 7 | 7
score on a scale | 9.71 (8.65) | 4.43 (4.50)

3. Primary Outcome: Target Behaviors (Caregivers)
Description: This measure captures the top 3 dementia behaviors exhibited by the PLWD and chosen by the caregiver to work on in the COPE program. At baseline, the caregiver selects and ranks the top 3 behaviors (assessed via the Neuropsychiatric Inventory brief questionnaire) and/or activities (assessed via the Caregiver Assessment of Function and Upset Function) and rates confidence levels (0 = not at all, 4 = extremely). Caregivers reassess confidence levels at the 4-month follow up. The means reported are the change scores from baseline to follow up. A positive value indicates greater confidence and a better outcome.
Time Frame: Baseline, 4 months
Population: 1 caregiver in the control group refused to complete the assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers Receiving COPE From Instructor-trained COPE Clinicians | Caregivers Receiving COPE From Module-trained COPE Clinicians
Number analyzed (Participants) | 6 | 7
score on a scale
  PLWD behavior ranked #1 in upset level by Caregiver | -0.33 (0.82) | 1.43 (0.79)
  PLWD behavior ranked #2 in upset level by Caregiver | 0.67 (1.63) | 1.00 (1.29)
  PLWD behavior ranked #3 in upset level by Caregiver | 0.60 (1.52) | 0.29 (1.11)

4. Secondary Outcome: Neuropsychiatric Inventory Brief Questionnaire (NPI-Q) (PLWDs)
Description: Presence of 12 neuropsychiatric symptoms related to dementia. Caregivers answer yes or no to behaviors exhibited by the PLWD in the month prior to enrollment.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | PLWDs Receiving COPE From Instructor-trained COPE Clinicians | PLWDs Receiving COPE From Module-trained COPE Clinicians
Number analyzed (Participants) | 7 | 7
Participants
  Delusions | 3 | 4
  Hallucinations | 2 | 3
  Agitation/Aggression | 5 | 6
  Depression | 3 | 5
  Anxiety | 6 | 6
  Elation/Europhia | 3 | 0
  Apathy/Indifference | 4 | 6
  Disinhibition | 3 | 4
  Irritability/Lability | 6 | 6
  Motor Disturbance | 3 | 3
  Nighttime behaviors | 5 | 7
  Appetite Change | 4 | 6

5. Secondary Outcome: Caregiver Assessment of Function and Upset Function (CAFU) (Caregivers)
Description: Caregivers report instrumental activities of daily living (IADLs) and activities of daily living (ADLs) support for PLWDs and their upset and confidence in providing support. CG chooses up to 16 IADLs/ADLs for which they provide support for the PLWD. Then, the CG rates their own upset level 0 (not upset) to 10 (extremely upset) and confidence level from 0 (not confident at all) to 10 (extremely confident) for each IADL/ADL. Upset and confidence scores are sums of 16 items rated 0-10 on Likert scale. Higher numbers for upset are negative and higher numbers for confidence are positive.
Time Frame: Baseline
Population: Caregivers report IADL and ADL support for PLWDs and their upset and confidence in providing support.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers Receiving COPE From Instructor-trained COPE Clinicians | Caregivers Receiving COPE From Module-trained COPE Clinicians
Number analyzed (Participants) | 7 | 7
score on a scale
  Report of ADL/IADLs | 8.00 (3.37) | 10.57 (2.88)
  Level of CG confidence for ADL/IADLs support (sum across 16 items on Likert scale 0-10): number analyzed (Participants) | 6 | 7
  Level of CG confidence for ADL/IADLs support (sum across 16 items on Likert scale 0-10) | 77.50 (32.17) | 100.7 (37.18)
  Level of CG upset for ADL/IADLs support (sum across 16 items on Likert scale 0-10) | 22.57 (8.38) | 22.43 (9.98)

6. Secondary Outcome: Zarit Burden Scale
Description: The Zarit Burden Scale (Short 12-items) measures caregiver burden via 12 items assessed via the caregiver as (0 = never, 5 = nearly always). Total scores range from 0 to 48 and indicate no to mild burden (0-10), mild to moderate burden (10-20) and high burden (> 20).
Time Frame: Baseline, 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers Receiving COPE From Instructor-trained COPE Clinicians | Caregivers Receiving COPE From Module-trained COPE Clinicians
Number analyzed (Participants) | 7 | 7
score on a scale | 16.71 (6.32) | 20.86 (11.68)

7. Secondary Outcome: Short Sense of Competence Questionnaire (SSCQ) (Caregivers)
Description: The 7-item SSCQ assesses CG sense of capability and confidence in providing assistance to relatives. Respondents respond to statements about being a caregiver on a 5-point Likert-type scale (1 = strongly agree, 2 = agree, 3 = neither agree not disagree, 4 = disagree, 5 = strongly disagree). Total scores at one time point range from 7-35. The SSCQ has demonstrated reliability (α=.76), content validity via expert consensus panel, and construct validity (r=.88).
Time Frame: Baseline, 4 months
Population: Participant data is missing for 1 caregiver in the control group as this participant refused to complete this measure at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers Receiving COPE From Instructor-trained COPE Clinicians | Caregivers Receiving COPE From Module-trained COPE Clinicians
Number analyzed (Participants) | 6 | 7
score on a scale | -0.17 (5.19) | 2.43 (2.99)

8. Secondary Outcome: Quality of Life in Alzheimer's Disease (QOL-AD) (PLWDs)
Description: Caregivers complete this 13-item questionnaire as proxies to measure the quality of life of the person living with dementia (PLWD). Points are assigned to each item (poor = 1, fair = 2, good = 3, excellent = 4). The total score is the sum of all 13 items that generates summary scales for physical components (PCS) and for mental health components (MCS). Total scores range from 13-52.
Time Frame: Baseline, 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PLWDs Receiving COPE From Instructor-trained COPE Clinicians | PLWDs Receiving COPE From Module-trained COPE Clinicians
Number analyzed (Participants) | 7 | 7
score on a scale | -1.71 (4.92) | -0.43 (4.69)

9. Secondary Outcome: Lubben Social Network Scale (LSNS) (Caregivers)
Description: Self-report measure of social engagement including family and friends via 12 items. Items assess how many people participant sees at different time periods (0 = none, 5 = nine of more) and how often participant has social interactions (0 = less than monthly, 5 = daily). Total scores range from 0 - 60.
Time Frame: Baseline
Population: One caregiver in the control group refused to answer this baseline measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers Receiving COPE From Instructor-trained COPE Clinicians | Caregivers Receiving COPE From Module-trained COPE Clinicians
Number analyzed (Participants) | 6 | 7
score on a scale | 35.33 (7.81) | 35.14 (3.44)

ADVERSE EVENTS:
Time Frame: 14 months
Groups:
- Instructor-trained COPE Clinicians: Clinicians from PACE sites randomized to this study arm (control) will receive instructor-led training in the evidence-based dementia care program called COPE and then deliver COPE to dyads at their site.
- COPE Module-trained Clinicians: Clinicians from PACE sites randomized to this study arm (intervention) will receive self-paced online module training in the evidence-based dementia care program called COPE and then deliver COPE to dyads at their site.
- Caregivers Receiving COPE From Module-trained COPE Clinicians: Caregivers of eligible PLWDS enrolled at PACE sites randomized to the intervention arm will be recruited by "module-trained COPE clinicians." After initial recruitment, the study team will carry out consent and screening procedures with caregivers and collect caregiver outcome data at baseline (before meeting with COPE clinicians) and follow-up (4 months post-implementation). Caregivers must complete a minimal dose of 4 sessions out of 10 to be included in follow-up measures. Outcomes will be reviewed for change from baseline to follow-up and compared to "caregivers receiving COPE from instructor-trained COPE clinicians" for non-inferiority.
  Care of Older Persons in their Environment (COPE) online module training: An online module version of training for clinicians (OTs and RNs) in the evidence-based dementia caregiving program called Care of Older Persons in their Environment (COPE) is the intervention being tested for non-inferiority against the usual instructor-led COPE training.
Arm/Group | Instructor-trained COPE Clinicians | COPE Module-trained Clinicians | Caregivers Receiving COPE From Instructor-trained COPE Clinicians | Caregivers Receiving COPE From Module-trained COPE Clinicians | PLWDs Receiving COPE From Instructor-trained COPE Clinicians | PLWDs Receiving COPE From Module-trained COPE Clinicians
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/7 | 0/7 | 2/7 | 2/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/7 | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/7 | 0/7 | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT04165213/Prot_SAP_000.pdf